CLINICAL TRIAL: NCT00528554
Title: Laser Acupuncture to Alleviate Nausea and Vomiting in Children and Adolescents Receiving Highly Emetogenic Chemotherapy. A Prospective, Double-Blinded, Placebo-Controlled Clinical Trial
Brief Title: Laser Acupuncture Against Nausea in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Children Hospital Homburg (Other)
Collaborators: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SG-07-HT-01
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-09

CONDITIONS: Nausea; Vomiting; Cancer
Keywords: CINV; chemotherapy induced nausea and vomiting (CINV)
MeSH Terms: conditions — Nausea; Vomiting; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Active laser acupuncture
  Interventions: Procedure: laser acupuncture
- B (Placebo Comparator): Placebo laser acupuncture
  Interventions: Procedure: placebo laser acupuncture

INTERVENTIONS:
Procedure: laser acupuncture — laser acupuncture according to traditional chinese medicine criteria, energy dosage 1J/point, average of 8 points to be treated, once daily during chemotherapy course
  Other Names: Laser device: Modulas handy 2/99, 830 nm continuous wave, 30 mv 3,8 W/cm2, schwamedico, Ehringshausen, Germany
  Arms: A
Procedure: placebo laser acupuncture — laser acupuncture according to traditional chinese medicine criteria, average of 8 points to be treated, once daily during chemotherapy course
  Other Names: placebo laser, Modulas Handy 2/99, schwamedico, Ehringshausen, Germany
  Arms: B

SUMMARY:
To investigate whether nonthermal low level laser acupuncture has beneficial effects on nausea and vomiting in children receiving highly emetogenic chemotherapy for a malignant solid tumor. In a previous crossover study comparing needle acupuncture to no intervention in an otherwise similar setting we found beneficial effects, but this trial was not even single-blinded and therefore the results are questionable. The hypothesis is that active laser acupuncture is more effective than placebo laser acupuncture concerning episodes of retching/vomiting (primary outcome measure) and rescue antiemetic medication (secondary outcome measure) with a fix standard antiemetic medication

ELIGIBILITY:
Inclusion Criteria:

* Age 0-17,
* Highly emetogenic chemotherapy with at least 4 similar courses of chemotherapy concerning applied drugs (equivalent dosages)

Exclusion Criteria:

* Age older than 17 years,
* Participation in another clinical trial on supportive care

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2007-09; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
episodes of retching/vomiting per day during 1 chemotherapy course | 1 chemotherapy course (5 days)

SECONDARY OUTCOMES:
rescue antiemetic medication during 1 chemotherapy course | 1 chemotherapy course (5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Gottschling, MD, Principal Investigator — University Children's Hospital Homburg, Germany; Norbert Graf, MD, PhD, Study Director — University Children's Hospital Homburg, Germany
Locations (2):
- Germany (2):
  - University Children's Hospital Tübingen, Tübingen, Baden-Wurttemberg
  - University Children's Hospital Homburg, Homburg, Saarland